CLINICAL TRIAL: NCT04849676
Title: Exploring the Effects of Neurofeedback on Spasticity and Motor Function in Individuals With Subacute and Chronic Incomplete Spinal Cord Injury
Brief Title: Neurofeedback to Improve Spasticity After Incomplete Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN20NE696; 288894 (Other: Integrated Research Application System)
Record Dates: First submitted 2021-04-15; First posted 2021-04-19 (Actual); Last update posted 2022-04-18 (Actual); Status verified 2022-04

CONDITIONS: Incomplete Spinal Cord Injury

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Upper limb subacute spinal cord injury (sUL) (Experimental): Intervention: neurofeedback. Participants will receive visual feedback on a screen.
  Diagnostic Tests:
  Modified Ashworth Scale grading muscle resistance to movement (all limbs tested)
  Perceived Spasticity level questionnaire on impact of spasticity
  Spinal Cord Independence Measure questionnaire on level of independence of patients
  Diary of spastic episodes
  Grip strength - measure of hand and forearm muscle strength using dynamometer
  Instrumented Pendulum test - oscillations when forearm is dropped from a resting position
  Hand grip - closing and opening the fist recorded with Kinect (Microsoft) device
  EEG recording in relaxed state with bioamplifier g.usbamp (Guger Technologies, Austria)
  Brief Visual Analog Scale self-assessment of performance and mental strategies
  Motor evoked potential - effect of therapy on the descending path from brain to spinal cord with a transcranial magnetic stimulator (200-2, Magstim Co Ltd)
  Interventions: Other: visual neurofeedback
- Upper limb chronic spinal cord injury (sUL) (Experimental): Intervention: neurofeedback. Participants will receive visual feedback on a screen.
  Diagnostic Tests:
  Modified Ashworth Scale grading muscle resistance to movement (all limbs tested)
  Perceived Spasticity level questionnaire on impact of spasticity
  Spinal Cord Independence Measure questionnaire on level of independence of patients
  Diary of spastic episodes
  Grip strength - measure of hand and forearm muscle strength using dynamometer
  Instrumented Pendulum test - oscillations when forearm is dropped from a resting position
  Hand grip - closing and opening the fist recorded with Kinect (Microsoft) device
  EEG recording in relaxed state with bioamplifier g.usbamp (Guger Technologies, Austria)
  Brief Visual Analog Scale self-assessment of performance and mental strategies
  Motor evoked potential - effect of therapy on the descending path from brain to spinal cord with a transcranial magnetic stimulator (200-2, Magstim Co Ltd)
  Interventions: Other: visual neurofeedback
- Lower limb subacute spinal cord injury (sLL) (Experimental): Intervention: neurofeedback. Participants will receive visual feedback on a screen.
  Diagnostic Tests:
  Modified Ashworth Scale grading muscle resistance to movement (all limbs tested)
  Perceived Spasticity level questionnaire on impact of spasticity
  Spinal Cord Independence Measure questionnaire on level of independence of patients
  Diary of spastic episodes
  Instrumented Pendulum test - oscillations when lower leg is dropped from a resting position
  10m walking test - patient walks 10 meters in a straight line, recorded with Kinect (Microsoft) device
  EEG recording in relaxed state with bioamplifier g.usbamp (Guger Technologies, Austria)
  Brief Visual Analog Scale self-assessment of performance and mental strategies
  Motor evoked potential - effect of therapy on the descending path from brain to spinal cord with a transcranial magnetic stimulator (200-2, Magstim Co Ltd)
  Interventions: Other: visual neurofeedback
- Lower limb chronic spinal cord injury (cLL) (Experimental): Intervention: neurofeedback. Participants will receive visual feedback on a screen.
  Diagnostic Tests:
  Modified Ashworth Scale grading muscle resistance to movement (all limbs tested)
  Perceived Spasticity level questionnaire on impact of spasticity
  Spinal Cord Independence Measure questionnaire on level of independence of patients
  Diary of spastic episodes
  Instrumented Pendulum test - oscillations when lower leg is dropped from a resting position
  10m walking test - patient walks 10 meters in a straight line, recorded with Kinect (Microsoft) device
  EEG recording in relaxed state with bioamplifier g.usbamp (Guger Technologies, Austria)
  Brief Visual Analog Scale self-assessment of performance and mental strategies
  Motor evoked potential - effect of therapy on the descending path from brain to spinal cord with a transcranial magnetic stimulator (200-2, Magstim Co Ltd)
  Interventions: Other: visual neurofeedback

INTERVENTIONS:
Other: visual neurofeedback — Neurofeedback is a neuromodulatory intervention that does not require applying external stimuli. It relies on displaying participants' brain activity in real time, with the aim of modifying it. Electrical activity (EEG) will be recorded from participants and displayed in real time on a computer screen, in the form of three bars. They will be asked to increase the middle bar, while keeping the side bars low.
  The intervention requires training to achieve voluntary control of the targeted brain activity.

SUMMARY:
After incomplete spinal cord injury (iSCI), many people still have control over their upper and/or lower limbs, but secondary conditions such as spasticity impair the function they have left. Spasticity includes increased reflex response and muscle tone, and is often painful. In this study we want to test a rehabilitation therapy to reduce spasticity after iSCI and improve participants' control over their extremities. The study involves recording participants' brain signals (EEG) and displaying them on a computer, so that they learn to control specific features derived from their brain waves. This is called neurofeedback (NF). Two studies conducted in our group that explored NF effect on central neuropathic pain in iSCI reported as incidental finding a decrease in spasms, muscle tightness and foot drop.

The effect of NF is immediate and lasts up to 24 hours. In this study, we will explore systematically the short- and medium-term effect of NF on a larger number of iSCI, to inform a potential randomized clinical trial.

Gaining control over one's brain activity requires practice and 80-90% people eventually learn the skill. Each participant will therefore attend five sessions of NF taking no longer than two hours each.

20 participants will be recruited and assigned to either upper or lower limb spasticity groups. This will allow us to determine if the mechanism of NF differs between arms and legs. Participants will be further grouped into sub-acute and chronic groups, depending on the time since injury, to pinpoint at what stage post-injury NF is the most effective.

All groups will receive the same number of NF sessions. The primary outcome of this study is the change in spasticity of the hand or leg, as measured by the Modified Ashworth Scale (MAS). Secondary outcomes include use of arm/leg, quality of life, and the relation between functional improvement and EEG changes. Outcomes will be compared before/after each session, and before/after the whole intervention period, both inter- and intra-group.

DETAILED DESCRIPTION:
The proposed study is a pilot exploratory study. It will be carried out on 20 chronic and sub-acute incomplete spinal cord injury participants who will receive five sessions of neurofeedback treatment, over two weeks. The duration and number of sessions is based on previous studies in which participants learned neurofeedback strategies after two practice sessions.

People who decide to take part will be assigned to one of the following groups: subacute lower limb (sLL), subacute upper limb (sUL), chronic lower limb (cLL) or chronic - upper limb (cUL). We will use existing clinical American Spinal Injury Association (ASIA) testing information to assess the level and completeness of injury, i.e. we will gain this information from patient notes following assessment performed by the healthcare professional.

The groups will undergo similar therapy sessions. The intervention comprises the same task - neurofeedback, or modulation of brain oscillations. However, the location of modulation will differ between UL and LL groups because different parts of the brain are responsible for arm and leg function. Participants in the subacute groups (sUL, sLL) will attend two additional assessments as their baseline condition might change from week to week. Due to the nature of exploratory studies, the assessments presented for each group are necessary to determine accurately the effect of neurofeedback on motor function. Therefore, assessments presented for each session are compulsory.

The subjects will receive the intervention therapy independent of any routine therapy session at Queen Elizabeth National Spinal Injuries Unit (QENSIU). The sessions will occur within the same 2-hour time window, as much as possible, to prevent normal diurnal variation in biophysical parameters (brain signatures, spasms).

Recruitment: The total number of patients admitted to the QENSIU with incomplete injury in 2019-20 was 105, comprising 69 cervical level (C1-C8), 22 thoracic level (T1-T12) and 13 lumbar level (L1-L5) with a mean length of stay of 38 days (5 weeks). The out-patient activity of the Unit: in 2019-20, 1551 individuals returned for post-discharge management of their injury and 70 new outpatients were accepted.

The total number of patients graded with an ASIA impairment level C or D in 2019/20 was: C = 29, D = 63, indicating that we should be able to recruit 10 participants with subacute SCI and 10 with chronic SCI over a period of 2 years. This number would allow us to perform non-parametric statistical analysis and to collect data that would inform power analysis for a future randomised controlled trail.

Patients will be identified and approached by their clinical consultants (Co-Investigator Dr. Mariel Purcell). Prior to participating, patients will be given information sheets and consent forms to sign. Should the participant themselves be physically unable to sign, a witnessed proxy will do so on the patient's behalf.

Assessments:

All participants will be assessed before, during and after the therapy as detailed below.

1. Pre- and post-therapy assessments Subacute SCI groups (sUL, sLL) will undergo two assessments before and two after the therapy period. The first and last assessments will take place one week before starting and one week after completing the NF sessions, respectively, to monitor changes in their baseline condition. Chronic participants (cUL, cLL) are considered stable, therefore only one pre- and one post-therapy assessment are needed. These will take place on the days of the first and last NF session, respectively.

   The pre-treatment and post-treatment assessments are identical and include the following tests:

   Everyone:
   1. Modified Ashworth Scale (MAS) grades the resistance of the muscle while the researcher moves the tested limb to full extension. Upper and lower limbs will be tested for both groups, to verify whether NF only affects spasticity in the targeted limbs, or its effect is general.
   2. Perceived Spasticity level (SCI-SET): participants assess the impact of spasticity during the past 7 days on 35 different items from -3 (extremely problematic) to +3 (extremely helpful).
   3. Spinal Cord Independence Measure (SCIM) questionnaire with the emphasis on the set of questions relevant for the use of the arms or legs.
   4. Diary of spastic episodes - all participants will keep a diary of daily spastic episodes starting a week before and ending a week after treatment.

      Lower limb groups (sLL and cLL) tests:
   5. Instrumented Pendulum test for lower limb to evaluate the level of thigh spasticity. A digital goniometer is placed on the participant's knee and the lower leg is dropped from a resting horizontal position, to observe the number and size of oscillations performed before stopping.
   6. Ten-meter walking test (10MWT) to assess the initial level of locomotion of the participant, and the impact of spasticity on walking. A motion recording device will be used to evaluate walking symmetry while the participant walks 10m in a straight line. The test may be video recorded in participants who consent to this option. This test only applies to participants who can walk (with or without assistance).

      Upper limb groups (sUL and cUL) tests:
   7. Grip strength (GS) test to measure the muscle strength of the hand and forearm with the help of a dynamometer. The participant will squeeze the dynamometer three times with each hand. GS only applies to participants who are able to flex their hand.
   8. Instrumented Pendulum test for upper limb (elbow), similar to (e).
   9. Hand grip - the participant will be asked to close and open their fist. A motion recording device will be used to evaluate hand function. This will be video recorded in participants who consent to it. Hand grip motion recording only applies to participants who are able to flex their hand.
2. Therapy The participants will receive 5 sessions of neurofeedback, delivered over two weeks. Interim assessments will be carried out at the beginning and end of each session.

2.1 Intervention One intervention session comprises five trials of visual neurofeedback, lasting 5 minutes each. Participants will receive visual feedback on a screen in the form of three bars that represent brain features, and will focus on modulating the central bar (alpha wave). The side bars are used to reduce signal noise from blinking and movement. All participants will perform the same task.

2.2 Interim assessments During the first two sessions, the participants can explore different strategies to control their brain activity. Changes in spasticity are expected after the third session, therefore the last three interim assessments include additional tests. Interim assessments for the first two sessions will take 35 minutes in total. Assessments performed during the last three sessions will take 70 minutes in total. Overall, sessions 3, 4 and 5 will take up to 2 hours each, including comfort breaks.

1. Baseline brain activity (EEG) will be recorded before and after each session. (everyone)
2. Recording of participants opening and closing their fist (sUL and cUL groups) before and after each session, using the motion sensing device.
3. 10-meter walking test (sLL and cLL groups) before and after each session. The test will be recorded using a motion sensing device.
4. Instrumented pendulum test (everyone) before and after the last three sessions, performed using a motion sensing device.
5. Modified Ashworth scale (everyone) before and after each session on selected upper or lower limb joints.
6. Brief Visual Analog Scale (VAS) self-assessment of performance and mental strategies after each session. (everyone)
7. Motor evoked potential (MEP) before and after the last three sessions, to determine the effect of the therapy on the descending path from the brain to the spinal cord. To obtain the MEP, a magnetic coil will be held above the participant's head and magnetic pulses will be applied. (everyone)

All equipment used in this study that is in direct contact with participants has medical device grade Certificate Europe (CE) mark.

EEG will be recorded with a g.Tech biosignal USB amplifier (Guger Technologies, Austria) which enables on-line EEG measurement, signal analysis and visualisation of EEG signals on a computer screen.

In summary, the first two sessions comprising the intervention and tests will take approximately 1 hour, and the last three sessions, which include additional assessments will last 2 hours, including comfort breaks. The five sessions will be completed within 2 weeks.

During the first assessment, patients will get advice and assistance from researchers when completing the questionnaires. For the second assessment they will be able to fill them out at home on their own.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for subacute upper limb:

1. Aged above 18
2. Incomplete injury to the spinal cord, resulting in ASIA level C or D SCI
3. Injury occurred no more than six months prior to participation in the study
4. Injury level C3 to C7
5. Normal or corrected to normal vision
6. Spasticity equivalent of MAS level 1+ and above

Inclusion Criteria for chronic upper limb:

1. Aged above 18
2. Incomplete injury to the spinal cord, resulting in ASIA level C or D SCI
3. Injury occurred more than one year prior to participation in the study
4. Injury level C3 to C7
5. Normal or corrected to normal vision
6. Spasticity equivalent of MAS level 1+ and above
7. Live in Greater Glasgow and Clyde area

Inclusion Criteria for subacute lower limb:

1. Aged above 18
2. Incomplete injury to the spinal cord, resulting in ASIA level C or D SCI
3. Injury occurred no more than six months prior to participation in the study
4. Injury level T1 to L1
5. Normal or corrected to normal vision
6. Ability to walk > 10 meters (assisted or unassisted), if ASIA level D
7. Spasticity equivalent of MAS level 1+ and above

Inclusion Criteria for chronic lower limb:

1. Aged above 18
2. Incomplete injury to the spinal cord, resulting in ASIA level C or D SCI
3. Injury occurred more than one year prior to participation in the study
4. Injury level T1 to L1
5. Normal or corrected to normal vision
6. Ability to walk > 10 meters (assisted or unassisted), if ASIA level D
7. Spasticity equivalent of MAS level 1+ and above
8. Live in Greater Glasgow and Clyde area

Exclusion Criteria:

Exclusion Criteria for subacute groups:

1. Participation in any other neurofeedback intervention group
2. Inability to understand the task
3. Self-reported neurological disorders e.g. previously confirmed peripheral nerve injury or brain injury
4. General poor health due to secondary consequences of injury
5. Conditions contra-indicative of neurostimulator usage (implanted devices, sensitive skin sores in the upper and lower extremities, pregnancy, severe autonomic dysreflexia)
6. History of epilepsy
7. Inability to sit for 1.5 hours
8. Inability to speak and/or understand English

Exclusion Criteria for chronic groups:

1. Participation in any other neurofeedback intervention group
2. Inability to understand the task
3. Self-reported neurological disorders e.g. previously confirmed peripheral nerve injury or brain injury
4. General poor health due to secondary consequences of injury
5. Conditions contra-indicative of neurostimulator usage (implanted devices, sensitive skin sores in the upper and lower extremities, pregnancy, severe autonomic dysreflexia)
6. History of epilepsy
7. Inability to sit for 1.5 hours
8. Inability to speak and/or understand English
9. Live outside Greater Glasgow and Clyde area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | 4 weeks
  Improvements in spasticity in the upper or lower limb (UL, LL groups) after neurofeedback sessions

SECONDARY OUTCOMES:
Functional improvements | 4 weeks
  Quantitative assessment of any functional improvements in the arms or legs
Participant experience | 1 hour; after the last experimental session
  Quantitative and qualitative analysis of participant experience and changes in quality of life
Correlation between EEG activity and functional improvements | one day to one month after the last experimental session, off line quantitative analysis
  To understand the relation between change in brain signatures as a result of neurofeedback, and improvements in arm or leg function, with the aim of describing neurofeedback mechanisms.

CONTACTS AND LOCATIONS:
Overall Officials: Mariel Purcell, MD, Principal Investigator — NHS Greater Galsgow and Clyde
Locations (1):
- Queen Elizabeth University Hospital, Queen Elizabeth National Spinal Injurie Unit, Glasgow, Glasgow City, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Shared on request
Supporting Information: Study Protocol
Time Frame: After study end (March 2023)
Access Criteria: Data will be shared upon reasonable request